CLINICAL TRIAL: NCT06552897
Title: A Randomized Controlled Trial Investigating the Efficacy of Combined Adductor Canal and Tibial Nerve Blocks for Enhanced Postoperative Pain Management in Knee Arthroplasty
Brief Title: Efficacy of Combined Adductor and Tibial Nerve Blocks for Pain Management in Knee Arthroplasty
Acronym: CATNAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, semih başkan, Associate Professor Dr. Semih Başkan, Department of Anesthesiology and Reanimation, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUACHT-2024-KA01
Record Dates: First submitted 2024-08-05; First posted 2024-08-14 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Pain Management; Total Knee Arthroplasty; Regional Anesthesia; Nerve Blocks
Keywords: Total knee arthroplasty; Adductor canal block,; Selective tibial nerve block; Postoperative analgesia,

STUDY DESIGN:
Intervention Model Description: This study uses a Parallel Assignment design in which participants undergoing total knee arthroplasty (TKA) are randomly assigned to one of two intervention groups.
  Group A: Receives an Adductor Canal Block (ACB) alone, which targets the nerves supplying the front and inner parts of the knee.
  Group AT: Receives a combination of Adductor Canal Block (ACB) and Selective Tibial Nerve Block (STNB), providing additional analgesia to the back of the knee.
  Both groups are assessed for postoperative pain relief, opioid consumption, side effects, and overall patient satisfaction. The parallel assignment allows for a direct comparison of the effectiveness and safety of these two pain management strategies.
Who Masked: Participant, Investigator
Masking Description: Double-blind (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Adductor Canal Block (ACB) Group, Arm 2: Combined Adductor Canal Block and Selective Tibial N (Other): Arm 1: Adductor Canal Block (ACB) Group Arm Type: Active Comparator Description: This group receives the standard intervention of an Adductor Canal Block (ACB), which serves as the control or comparator arm in the study.
  Interventions: Procedure: Intervention 1: Adductor Canal Block (ACB)
- Arm 2: Combined Adductor Canal Block and Selective Tibial Nerve Block (ACB + STNB) Group (Other): Arm 2: Combined Adductor Canal Block and Selective Tibial Nerve Block (ACB + STNB) Group Arm Type: Experimental Description: This group receives the experimental intervention combining Adductor Canal Block (ACB) with Selective Tibial Nerve Block (STNB) to evaluate its efficacy in enhancing postoperative analgesia.
  Interventions: Procedure: Intervention 2: Combined Adductor Canal Block and Selective Tibial Nerve Block (ACB + STNB)

INTERVENTIONS:
Procedure: Intervention 1: Adductor Canal Block (ACB) — For the Interventions section, you should describe the specific procedures or treatments administered in each arm of your study. Here's how you might present the interventions:
  Intervention 1: Adductor Canal Block (ACB) Name: Adductor Canal Block (ACB) Type: Procedure
  Description:
  Participants receive an ultrasound-guided adductor canal block. Dose and Administration: 20 ml of 0.25% bupivacaine is injected to target the saphenous nerve within the adductor canal.
  Objective: To provide analgesia to the anterior and medial aspects of the knee, preserving motor function to facilitate early mobilization.
  Arms: Arm 1: Adductor Canal Block (ACB) Group, Arm 2: Combined Adductor Canal Block and Selective Tibial N
Procedure: Intervention 2: Combined Adductor Canal Block and Selective Tibial Nerve Block (ACB + STNB) — Name: Combined Adductor Canal Block and Selective Tibial Nerve Block (ACB + STNB) Type: Procedure
  Description:
  Participants receive an ultrasound-guided adductor canal block followed by a selective tibial nerve block.
  Dose and Administration:
  Adductor Canal Block (ACB): 20 ml of 0.25% bupivacaine. Selective Tibial Nerve Block (STNB): 20 ml of 0.25% bupivacaine. Objective: To provide comprehensive analgesia to both the anterior and posterior aspects of the knee, aiming to enhance pain relief and reduce opioid consumption.
  Arms: Arm 2: Combined Adductor Canal Block and Selective Tibial Nerve Block (ACB + STNB) Group

SUMMARY:
This study aims to explore methods for enhancing pain relief following knee replacement surgery, a prevalent procedure for individuals with severe knee arthritis. Effective postoperative pain management is essential for ensuring a swift and comfortable recovery. Traditional pain management methods often involve medications that may have side effects; therefore, this study examines alternative approaches utilizing nerve blocks.

Two pain management methods are compared in this study:

Adductor Canal Block (ACB) Alone: A technique that numbs the anterior and medial regions of the knee.

Combined Adductor Canal Block and Selective Tibial Nerve Block (ACB + STNB): An innovative approach that includes an additional block to numb the posterior aspect of the knee.

The objective is to determine whether the combined approach offers superior pain relief, reduces the reliance on pain medications, and enhances overall postoperative recovery. Participants are randomly assigned to one of the two groups and receive the nerve blocks during their surgery.

This study aspires to contribute to the development of improved pain management strategies, facilitating quicker and more comfortable recovery for patients undergoing knee replacement surgery.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA), or knee replacement surgery, is a highly effective treatment for severe knee arthritis, providing significant pain relief and improved joint function. However, managing postoperative pain remains a significant challenge. Effective pain control is essential for facilitating early mobilization, reducing complications, and enhancing overall recovery.

Traditional pain management often relies heavily on opioids, which can cause side effects such as nausea, dizziness, and dependency. To address these concerns, regional anesthesia techniques, including nerve blocks, are increasingly utilized to provide targeted pain relief while minimizing opioid use.

This study evaluates the effectiveness of two nerve block techniques in managing postoperative pain following TKA:

Adductor Canal Block (ACB): This technique targets nerves in the adductor canal, primarily affecting the saphenous nerve, which provides sensation to the anterior and medial regions of the knee. ACB is recognized for preserving muscle strength, thereby facilitating early mobility.

Combined Adductor Canal Block and Selective Tibial Nerve Block (ACB + STNB): This approach incorporates a tibial nerve block to address the posterior aspect of the knee, aiming to provide comprehensive pain relief to both the anterior and posterior regions of the knee.

The study is a prospective, randomized controlled trial involving 76 patients undergoing TKA at Health Sciences University Ankara City Hospital. Participants are randomly assigned to receive either the ACB alone or the combined ACB + STNB.

Objectives:

To assess the effectiveness of the combined ACB + STNB in reducing postoperative pain compared to ACB alone.

To evaluate the impact on opioid consumption and overall patient satisfaction. To monitor potential side effects and the time to first additional analgesic requirement.

Methods:

Pain is measured using the Visual Analog Scale (VAS) at multiple time points after surgery.

The study also records total analgesic consumption via patient-controlled analgesia (PCA).

Secondary outcomes include side effects and patient satisfaction scores. The findings of this study could influence future pain management strategies for knee replacement surgeries, potentially offering patients a safer and more effective method for managing postoperative pain with fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

Age: 18 to 80 years. ASA Classification: Patients classified as ASA I, II, or III. Surgical Procedure: Scheduled for primary unilateral total knee arthroplasty (TKA) under combined spinal-epidural anesthesia.

Informed Consent: Ability to understand and provide written informed consent for participation in the study.

Exclusion Criteria:

ASA Classification: Patients classified as ASA IV or V. Surgical History: Revision TKA or any previous knee surgeries on the affected joint.

Medical Conditions:

Infection or neuropathy at the injection site. Coagulopathy or use of anticoagulant medications. Severe cardiac, hepatic, respiratory, or renal disease. Diagnosis of diabetic neuropathy. History of cerebrovascular accident with motor or sensory deficits. Neuropsychiatric disorders that affect cognition or communication.

Pain Management:

Inability to understand or use the Visual Analog Scale (VAS) for pain assessment.

Long-term use of analgesic therapy that could interfere with study assessments. Allergies: Known allergy to local anesthetics used in the study. Block Failure: Failed blocks or anesthesia issues prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Levels | Pain levels will be assessed at 0, 1, 2, 8, 12, and 24 hours following the completion of the surgical procedure.
  The intensity of postoperative pain will be evaluated using the Visual Analog Scale (VAS), a widely used pain assessment tool.Measurement Details: The VAS is a 10-point scale where 0 represents "no pain" and 10 represents "the worst pain imaginable." Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Total Analgesic Consumption | Within the first 24 hours post-surgery.
  Pain levels will be assessed at 0, 1, 2, 8, 12, and 24 hours following the completion of the surgical procedure.
Time to First Additional Analgesic Request | Within the first 24 hours post-surgery
  Description: The time elapsed from the end of surgery to the first request for additional analgesics will be recorded.
  Measurement Details: The time (in minutes) from the completion of surgery until the first patient-initiated request for additional analgesia will be measured. A longer duration indicates better initial pain control.
Incidence of Side Effects | Within the first 24 hours post-surgery.
  Description: The incidence of side effects such as nausea, vomiting, and hypotension will be documented.
  Measurement Details: The occurrence of these side effects will be recorded as a binary outcome (yes/no). Additionally, the severity of side effects will be assessed using standard clinical grading scales.
Patient Satisfaction | Assessed 24 hours post-surgery.
  Patient satisfaction regarding pain management and overall experience will be measured.
  Measurement Details: Satisfaction will be assessed using a 5-point Likert scale, where 1 represents "very dissatisfied" and 5 represents "very satisfied." Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Semih Başkan, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Health Sciences University Ankara City Hospital, Etimesgut, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Terkawi AS, Mavridis D, Sessler DI, Nunemaker MS, Doais KS, Terkawi RS, Terkawi YS, Petropoulou M, Nemergut EC. Pain Management Modalities after Total Knee Arthroplasty: A Network Meta-analysis of 170 Randomized Controlled Trials. Anesthesiology. 2017 May;126(5):923-937. doi: 10.1097/ALN.0000000000001607. PMID 28288050
- [Result] Jaeger P, Koscielniak-Nielsen ZJ, Schroder HM, Mathiesen O, Henningsen MH, Lund J, Jenstrup MT, Dahl JB. Adductor canal block for postoperative pain treatment after revision knee arthroplasty: a blinded, randomized, placebo-controlled study. PLoS One. 2014 Nov 11;9(11):e111951. doi: 10.1371/journal.pone.0111951. eCollection 2014. PMID 25386752
- [Result] Marty P, Chassery C, Rontes O, Vuillaume C, Basset B, Merouani M, Marquis C, De Lussy A, Ferre F, Naudin C, Joshi GP, Delbos A. Combined proximal or distal nerve blocks for postoperative analgesia after total knee arthroplasty: a randomised controlled trial. Br J Anaesth. 2022 Sep;129(3):427-434. doi: 10.1016/j.bja.2022.05.024. Epub 2022 Jun 28. PMID 35773028